CLINICAL TRIAL: NCT04141527
Title: Spinal Sufentanil for Relief of Labor Pain in Primi- and Multiparous Parturients
Brief Title: Spinal Sufentanil for Obstetric Analgesia
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: DNR2015/687
Record Dates: First submitted 2019-10-17; First posted 2019-10-28 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Labor Pain
Keywords: Labor; Intrathecal sufentanil; Obstetrical; Spinal analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primiparous women: 82 primiparous obstetrical patients given intrathecal sufentanil for labor pain.
  Interventions: Procedure: Spinal analgesia
- Multiparous women: 82 multiparous obstetrical patients given intrathecal sufentanil for labor pain.
  Interventions: Procedure: Spinal analgesia

INTERVENTIONS:
Procedure: Spinal analgesia — Spinal analgesia (SA) was provided by a resident or specialist anaesthesiologist with the patient in a sitting or a recumbent position. A pencil-point needle, primarily 27 G (0.4 mm), otherwise 25 G (0.5 mm), was used for transdermal intrathecal administration of 2.0 ml of sufentanil 5 µg/ml (Sufenta®, Janssen-Cilag AB, Solna, Sweden) at low-lumbar level. Blood pressure was recorded before, immediately after, and at five-minute intervals for 20 minutes after the block. Any decrease in systolic pressure to <100 mmHg or a decrease >20% from the baseline level despite infusion of crystalloid was defined to indicate maternal hypotension.

SUMMARY:
Background: This descriptive study was designed to evaluate effects and adverse effects of spinal sufentanil for relief of labor pain in primi- and multiparous women.

Methods: The retrospective study design was approved by the regional Human Research Ethics Review Board, Lund, Sweden (Dnr 2015/687). The investigators included 164 (82 primi- and 82 multiparous) obstetrical patients given 10 µg of intrathecal sufentanil for labor pain. Any maternal hypotension, third- or fourth-degree perineal tear, intrapartum Cesarean section, abnormal fetal heart rate, low Apgar score, use of neonatal intensive care, postdural puncture headache, epidural blood patch, and breastfeeding problem was recorded. Major outcome measures were maternal satisfaction with pain relief, and provision of supplementary analgesia.

DETAILED DESCRIPTION:
A total sample size of 150 parturients had been calculated to enable differences of at least 20 % versus 5.0 % in proportions of obstetrical and neonatal problems between (equal numbers of) primi- and multiparous mothers to be statistically confirmed with 80 % power and 95 % probability.

Descriptive parametric data is reported as mean ± standard deviation (SD), and descriptive non-parametric data as median with interquartile range (IQR). Proportions are reported in percent with 95 % confidence interval (CI).

Parametric data was compared with two-tailed unpaired student's t-test, and non-parametric data with the Mann-Whitney U-test. Proportions were analyzed with two-tailed Fisher's exact test.

Probability (P) values at < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Intrathecal sufentanil for labor pain

Exclusion Criteria:

Demographic, obstetrical or neonatal data is missing

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women in labor
Study Population: Primi- and multiparous obstetrical patients at the maternity ward of the Central Hospital in Kristianstad, Sweden, between 7th January 2013 and 29th July 2016
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Maternal hypotension | During the first 20 minutes after spinal analgesia with 5 minutes intervals
  Any fall in systolic pressure to <100 mmHg or a decrease >20% from the baseline level
Fetal bradycardia | During the first hour after spinal analgesia
  A decrease in FHR(fetal heart rate) to 80 beats/ min for duration of 2 or more
Late fetal deceleration | During the first hour after spinal analgesia
  FHR(fetal heart rate)<FHR 40 min beats/ min below the baseline or less than 90/beats min for duration of 2 minutes or more
Supplementary spinal analgesia | 24 hours after initial spinal analgesia
  Any use of spinal analgesia after primary spinal analgesia
Supplementary epidural analgesia | 24 hours after initial spinal analgesia
  Any use of epidural analgesia after primary spinal analgesia
Instrumental delivery | During childbirth
  Use of instrumental delivery
Intrapartum Cesarean section | During childbirth
  Use of intrapartum Cesarean section
Third- or fourth-degree perineal tear | During childbirth
  Rate of third- or fourth-degree perineal tear
Oxytocin before spinal analgesia | 24 hours before childbirth
  Any use of oxytocin before spinal analgesia
Oxytocin after spinal analgesia | 24 hours after spinal analgesia
  Any use of oxytocin after spinal analgesia
Maternal satisfaction with pain relief | 24 hours after spinal analgesia
  Defined by parturient after delivery as very god, god, less satisfactory or bad
Postspinal dural puncture headache | 48 hours after spinal analgesia
  Rate of postspinal dural puncture headache
Epidural blood patch | 1 veek after spinal analgesia
  Use of epidural blood patch

SECONDARY OUTCOMES:
Low Apgar score of newborn (Apgar score ≤ 7 ) | One minute and 5 minutes after birth
  Number of newborns with Apgar score ≤ 7
Use of neonatal intensive care | 1 week
  Number of newborns requiring intensive care unit
Breastfeeding | 1 week
  Number of infants with breastfeeding
Time from maternal arrival until request for SA | During childbirth
  Time in minutes
Time from request for SA until arrival of anaesthesiologist | During childbirth
  Time in minutes
Time from arrival of anaesthesiologist until SA | During childbirth
  Time in minutes
Time from SA until maximal cervical dilation | During childbirth
  Time in minutes
Time from maximal cervical dilation until delivery | During childbirth
  Time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Åkeson, Professor, Principal Investigator — Lund University Skåne University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Loubert C, Hinova A, Fernando R. Update on modern neuraxial analgesia in labour: a review of the literature of the last 5 years. Anaesthesia. 2011 Mar;66(3):191-212. doi: 10.1111/j.1365-2044.2010.06616.x. PMID 21320088
- [Background] Eriksson SL, Blomberg I, Olofsson C. Single-shot intrathecal sufentanil with bupivacaine in late labour--analgesic quality and obstetric outcome. Eur J Obstet Gynecol Reprod Biol. 2003 Oct 10;110(2):131-5. doi: 10.1016/s0301-2115(03)00049-6. PMID 12969571
- [Background] Campbell DC, Camann WR, Datta S. The addition of bupivacaine to intrathecal sufentanil for labor analgesia. Anesth Analg. 1995 Aug;81(2):305-9. doi: 10.1097/00000539-199508000-00017. PMID 7618720
- [Background] Sia AT, Chong JL, Chiu JW. Combination of intrathecal sufentanil 10 mug plus bupivacaine 2.5 mg for labor analgesia: is half the dose enough? Anesth Analg. 1999 Feb;88(2):362-6. doi: 10.1097/00000539-199902000-00026. PMID 9972757
- [Background] Aneiros F, Vazquez M, Valino C, Taboada M, Sabate S, Otero P, Costa J, Carceller J, Vazquez R, Diaz-Vieito M, Rodriguez A, Alvarez J. Does epidural versus combined spinal-epidural analgesia prolong labor and increase the risk of instrumental and cesarean delivery in nulliparous women? J Clin Anesth. 2009 Mar;21(2):94-7. doi: 10.1016/j.jclinane.2008.06.020. PMID 19329011
- [Background] Norris MC, Fogel ST, Conway-Long C. Combined spinal-epidural versus epidural labor analgesia. Anesthesiology. 2001 Oct;95(4):913-20. doi: 10.1097/00000542-200110000-00020. PMID 11605932
- [Background] Stocks GM, Hallworth SP, Fernando R, England AJ, Columb MO, Lyons G. Minimum local analgesic dose of intrathecal bupivacaine in labor and the effect of intrathecal fentanyl. Anesthesiology. 2001 Apr;94(4):593-8; discussion 5A. doi: 10.1097/00000542-200104000-00011. PMID 11379678
- [Background] Patel NP, Armstrong SL, Fernando R, Columb MO, Bray JK, Sodhi V, Lyons GR. Combined spinal epidural vs epidural labour analgesia: does initial intrathecal analgesia reduce the subsequent minimum local analgesic concentration of epidural bupivacaine? Anaesthesia. 2012 Jun;67(6):584-93. doi: 10.1111/j.1365-2044.2011.07045.x. Epub 2012 Mar 15. PMID 22420645
- [Background] Valensise H, Lo Presti D, Tiralongo GM, Pisani I, Gagliardi G, Vasapollo B, Frigo MG. Foetal heart rate deceleration with combined spinal-epidural analgesia during labour: a maternal haemodynamic cardiac study. J Matern Fetal Neonatal Med. 2016;29(12):1980-6. doi: 10.3109/14767058.2015.1072156. Epub 2015 Aug 28. PMID 26333691
- [Background] Patel NP, El-Wahab N, Fernando R, Wilson S, Robson SC, Columb MO, Lyons GR. Fetal effects of combined spinal-epidural vs epidural labour analgesia: a prospective, randomised double-blind study. Anaesthesia. 2014 May;69(5):458-67. doi: 10.1111/anae.12602. PMID 24738803
- [Background] Anim-Somuah M, Smyth R, Howell C. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD000331. doi: 10.1002/14651858.CD000331.pub2. PMID 16235275
- [Background] Laine K, Gissler M, Pirhonen J. Changing incidence of anal sphincter tears in four Nordic countries through the last decades. Eur J Obstet Gynecol Reprod Biol. 2009 Sep;146(1):71-5. doi: 10.1016/j.ejogrb.2009.04.033. Epub 2009 May 30. PMID 19482405
- [Background] Howell CJ, Kidd C, Roberts W, Upton P, Lucking L, Jones PW, Johanson RB. A randomised controlled trial of epidural compared with non-epidural analgesia in labour. BJOG. 2001 Jan;108(1):27-33. doi: 10.1111/j.1471-0528.2001.00012.x. PMID 11213000
- [Background] Cooper GM, MacArthur C, Wilson MJ, Moore PA, Shennan A; COMET Study Group UK. Satisfaction, control and pain relief: short- and long-term assessments in a randomised controlled trial of low-dose and traditional epidurals and a non-epidural comparison group. Int J Obstet Anesth. 2010 Jan;19(1):31-7. doi: 10.1016/j.ijoa.2009.05.004. Epub 2009 Nov 27. PMID 19945274
- [Background] Choi PT, Galinski SE, Takeuchi L, Lucas S, Tamayo C, Jadad AR. PDPH is a common complication of neuraxial blockade in parturients: a meta-analysis of obstetrical studies. Can J Anaesth. 2003 May;50(5):460-9. doi: 10.1007/BF03021057. PMID 12734154
- [Background] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Background] Van de Velde M, Schepers R, Berends N, Vandermeersch E, De Buck F. Ten years of experience with accidental dural puncture and post-dural puncture headache in a tertiary obstetric anaesthesia department. Int J Obstet Anesth. 2008 Oct;17(4):329-35. doi: 10.1016/j.ijoa.2007.04.009. Epub 2008 Aug 8. PMID 18691871
- [Background] Camann W, Abouleish A, Eisenach J, Hood D, Datta S. Intrathecal sufentanil and epidural bupivacaine for labor analgesia: dose-response of individual agents and in combination. Reg Anesth Pain Med. 1998 Sep-Oct;23(5):457-62. doi: 10.1016/s1098-7339(98)90027-x. PMID 9773697
- [Background] Clarke VT, Smiley RM, Finster M. Uterine hyperactivity after intrathecal injection of fentanyl for analgesia during labor: a cause of fetal bradycardia? Anesthesiology. 1994 Oct;81(4):1083. doi: 10.1097/00000542-199410000-00041. No abstract available. PMID 7943823
- [Background] Harsten A, Gillberg L, Hakansson L, Olsson M. Intrathecal sufentanil compared with epidural bupivacaine analgesia in labour. Eur J Anaesthesiol. 1997 Nov;14(6):642-5. doi: 10.1046/j.1365-2346.1994.00212.x. PMID 9466102
- [Result] Abouleish A, Abouleish E, Camann W. Combined spinal-epidural analgesia in advanced labour. Can J Anaesth. 1994 Jul;41(7):575-8. doi: 10.1007/BF03009995. PMID 8087904
- [Result] D'Angelo R, Anderson MT, Philip J, Eisenach JC. Intrathecal sufentanil compared to epidural bupivacaine for labor analgesia. Anesthesiology. 1994 Jun;80(6):1209-15. doi: 10.1097/00000542-199406000-00007. PMID 8010467
- [Result] Herman NL, Calicott R, Van Decar TK, Conlin G, Tilton J. Determination of the dose-response relationship for intrathecal sufentanil in laboring patients. Anesth Analg. 1997 Jun;84(6):1256-61. doi: 10.1097/00000539-199706000-00016. PMID 9174303
- [Result] Mardirosoff C, Dumont L, Boulvain M, Tramer MR. Fetal bradycardia due to intrathecal opioids for labour analgesia: a systematic review. BJOG. 2002 Mar;109(3):274-81. doi: 10.1111/j.1471-0528.2002.01380.x. PMID 11950182
- [Result] Everaert N, Coppens M, Vlerick P, Braems G, Wouters P, De Hert S. Combined spinal epidural analgesia for labor using sufentanil epidurally versus intrathecally: a retrospective study on the influence on fetal heart trace. J Perinat Med. 2015 Jul;43(4):481-4. doi: 10.1515/jpm-2014-0077. PMID 24922321
- [Result] Junttila EK, Karjalainen PK, Ohtonen PP, Raudaskoski TH, Ranta PO. A comparison of paracervical block with single-shot spinal for labour analgesia in multiparous women: a randomised controlled trial. Int J Obstet Anesth. 2009 Jan;18(1):15-21. doi: 10.1016/j.ijoa.2008.01.020. Epub 2008 Sep 26. PMID 18823774
- [Result] Wilson MJ, MacArthur C, Cooper GM, Bick D, Moore PA, Shennan A; COMET Study Group UK. Epidural analgesia and breastfeeding: a randomised controlled trial of epidural techniques with and without fentanyl and a non-epidural comparison group. Anaesthesia. 2010 Feb;65(2):145-53. doi: 10.1111/j.1365-2044.2009.06136.x. Epub 2009 Nov 12. PMID 19912160
- See also: Statistics on breastfeeding 2014. Statistics Sweden 2016 — http://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/statistik/2016-9-19.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT04141527/Prot_SAP_000.pdf